CLINICAL TRIAL: NCT04441697
Title: Monitoring of Sleepiness in Patients With Parkinson's Disease Before and During Treatment With Continuous Dopaminergic Delivery Device or Deep Brain Stimulation
Brief Title: Sleepiness in Parkinson's Patients With Continuous Dopaminergic Delivery Device or Deep Brain Stimulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI085
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
Keywords: continous dopaminergic delivery device; deep brain stimulation; sleepiness
MeSH Terms: conditions — Parkinson Disease; Sleepiness | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- continuous apomorphine delivery: apomorphine, subcutaneous administration, continuous delivery during 8 to 24 hours/day
  Interventions: Diagnostic Test: Multiple sleep latency tests
- continous levodopa/carbidopa delivery: levodopa/carbidopa monohydrate, jejunal administration, continuous delivery during 8 to 24 hours/day
  Interventions: Diagnostic Test: Multiple sleep latency tests
- deep brain stimulation: bilateral subthalamic electrical stimulation, intracranial neurosurgical electrodes, individual electrical parameters settings
  Interventions: Diagnostic Test: Multiple sleep latency tests

INTERVENTIONS:
Diagnostic Test: Multiple sleep latency tests — The investigators measure the objective sleepiness by recording the electro-encephalogramm during four experimental diurnal naps. They also perform a nocturnal polysomnography prior to the tests for a better interpretation.
  Other Names: Polysomnography

SUMMARY:
Sleepiness is frequent in parkinsonian patients, increasing with the duration of disease. By patients with motor fluctuations, continuous dopaminergic delivery devices or deep brain stimulation are justified to improve the motor prognosis. Antiparkinsonian treatments, especially dopaminergic agonists, may worsen the sleepiness and thus affect the quality of life. The investigators aimed to monitor sleepiness in parkinsonian patients before and during treatment with continous dopaminergic delivery device or deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* patient with Parkinson's disease and motor fluctuations
* and indicated for a continuous dopaminergic delivery device or deep brain stimulation

Exclusion Criteria:

* age < 18 years
* refusal for the continuous dopaminergic delivery device or deep brain stimulation
* wake-promoting drugs intake
* refusal to participate
* legal protection
* uncontrolled sleep apnea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients refered to the expert Parkinson Center of the Nancy University Hospital, with the diagnosis of Parkinson's disease at the stage of motor fluctuations, and indicated for a continuous dopaminergic delivery device or deep brain stimulation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Mean sleep latency | before continuous antiparkinsonian treatment
  Algebric mean (in minutes) of the sleep latency for the four experimental naps
Mean sleep latency | 6 months after continuous antiparkinsonian treatment
  Algebric mean (in minutes) of the sleep latency for the four experimental naps
Mean sleep latency | 12 months after continous antiparkinsonian treatment
  Algebric mean (in minutes) of the sleep latency for the four experimental naps

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi Siaghy, Study Chair — Research and Innovation Department
Locations (1):
- Nancy University Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No